CLINICAL TRIAL: NCT02075593
Title: ING200336: A Prospective, Interventional Pharmacokinetic and Safety Study of DTG/ABC/3TC in Pregnant Women
Brief Title: ING200336, Pharmacokinetic and Safety Study in Pregnant Women With Human Immuno Virus Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200336
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Results first posted 2022-02-18 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-08

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections; Arthralgia
Keywords: dolutegravir/abacavir/lamivudine fixed dose combination; pregnant women; once daily; antiretroviral therapy-naive; HIV-1 Infection; integrase inhibitor
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections; Arthralgia | interventions — dolutegravir; abacavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DTG/ABC/3TC (Experimental): All subjects will be administered DTG 50 milligrams (mg)/ABC 600 mg/3TC 300 mg FDC tablet once daily, with or without food.
  Interventions: Drug: DTG 50 mg /ABC 600 mg /3TC 300 mg FDC tablets

INTERVENTIONS:
Drug: DTG 50 mg /ABC 600 mg /3TC 300 mg FDC tablets — The DTG 50 mg /ABC 600 mg /3TC 300 mg FDC tablet is a purple, oval, biconvex tablets. The tablet contains 52.6 mg DTG sodium which is equivalent to 50 mg DTG free acid, 702 mg ABC sulphate which is equivalent to 600 mg ABC and 300 mg 3TC.

SUMMARY:
In this study, the dolutegravir/abacavir/lamivudine (DTG/ABC/3TC) fixed dose combination (FDC) tablet is being made available to women who become pregnant while participating in study ING117172. Continuation of antiretroviral therapy (ART) is key to both mother and the unborn fetus in order to maintain virologic suppression in the mother (thereby decreasing the risk for maternal disease progression), but also to reduce the risk of maternal-fetal transmission of human immunodeficiency virus type 1 (HIV-1) to her unborn child. This study also offers the first opportunity to investigate the impact of pregnancy on DTG pharmacokinetics (PK). This is an open-label, single arm interventional study. The number of women that will be enrolled into this study cannot be established a priori, as unintended pregnancies cannot be determined in advance. The maximum number of women would include all of those women randomized to DTG/ABC/3TC FDC (approximately 237), though unintended pregnancies in all of these women would not be anticipated.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected females participating in ING117172 on the DTG/ABC/3TC treatment arm who became pregnant with a singleton and have not met any safety or confirmed virologic withdrawal criteria.
* Signed and dated written informed consent is obtained from the subject or the subject's legal representative prior to screening.
* Willingness and intent to continue pregnancy
* Willingness to continue to receive DTG/ABC/3TC FDC.
* Willingness to enter the Antiretroviral Pregnancy Registry.
* Willingness to share medical information about herself and her infant for collection of delivery and infant outcomes as it relates to this study.
* Subjects enrolled in France: a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* History of allergy/sensitivity to DTG, ABC and/or 3TC.
* History of severe pre-clampsia, eclampsia, or hemolysis, elevated liver enzymes and low platelet count (HELLP)
* Any evidence of an active Center for Disease Control and Prevention (CDC) Category C disease, except cutaneous Kaposi's sarcoma not requiring systemic therapy or historic or current CD4+ cell levels <200 cells/millimeter^3.
* Subjects with any degree of hepatic impairment.
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical intraepithelial neoplasia; other localized malignancies require agreement between the investigator and the Study medical monitor for inclusion of the subject.
* Subjects who in the investigator's judgment, poses a significant suicidality risk. Recent history of suicidal behavior and/or suicidal ideation may be considered as evidence of serious suicide risk.
* Subjects with evidence of ongoing hepatitis B infection at screening, or anticipated need for Hepatitis C Virus therapy during the study.
* Treatment with any of the following agents within 28 days of Baseline: radiation therapy; cytotoxic chemotherapeutic agents; any immunomodulators that alter immune responses.
* Subjects enrolled in France: the subject has participated in any study using an investigational drug during the previous 60 days or 5 half-lives, or twice the duration of the biological effect of the experimental drug or vaccine, whichever is longer, prior to screening for the study or the subject will participate simultaneously in another clinical study.
* Any verified Grade 4 laboratory abnormality with the exception of Grade 4 lipid abnormalities (total cholesterol, triglycerides, high density lipoprotein [HDL] cholesterol, low density lipoprotein [LDL] cholesterol). A single repeat test is allowed during the Screening period to verify a result.
* Any acute laboratory abnormality observed in ING117172 or in any Screening laboratory assessments for ING200336, which, in the opinion of the Investigator, would preclude the subject's participation in the study.
* Hyperbilirubinemia of unknown etiology.
* Confirmed (with no more than 1 repeat evaluation) Grade >= 2 urine protein (dipstick), serum creatinine, total bilirubin, alanine aminotransferase or aspartate aminotransferase at the time of the screening lab.
* Subject has Creatinine Clearance of <50 mL/minute via Cockroft-Gault method at the time of the screening visit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-12-17 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2021-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (3):
- Russia (2):
  - GSK Investigational Site, Oryol
  - GSK Investigational Site, Saint Petersburg
- GSK Investigational Site, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a single arm open-label study in women who became pregnant while participating in study ING117172 (NCT01910402).
Pre-assignment Details: In this study, 4 pregnant women were enrolled. Participant flow data was collected only in pregnant women (enrolled population/study participants) and not in infants, as infants were not considered as enrolled per study design.
Groups:
- DTG/ABC/3TC - Mother: Participants (pregnant women) received fixed dose combination (FDC) tablet of dolutegravir (DTG) 50 milligrams (mg), abacavir (ABC) 600 mg and lamivudine (3TC) 300 mg once daily, with or without food.
Period: Overall Study
Arm/Group | DTG/ABC/3TC - Mother
Started | 4
Infants Born to Pregnant Women Who Received at Least One Dose of Study Treatment | 4
Completed | 3
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics data was collected only in pregnant women (enrolled population/study participants) and not in infants, as infants were not considered as enrolled per study design.
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.3 (5.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian/European heritage | 4

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Time Curve at Steady State During a Dosing Interval (AUC [0-tau]) for Dolutegravir
Description: Blood samples were collected at indicated timepoints for Pharmacokinetic (PK) analysis of dolutegravir at Trimester 2 (Weeks 18-26 of pregnancy), Trimester 3 (Weeks 30-36 of pregnancy) and at 8-12 Weeks postpartum.
Time Frame: Pre-dose and at 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose at Trimester 2 (Weeks 18-26 of pregnancy), Trimester 3 (Weeks 30-36 of pregnancy) and at 8-12 Weeks postpartum
Population: Pharmacokinetic Population consists of all participants in the Safety Population (comprised of all participants [pregnant women] who received at least one dose of study treatment) who had at least 1 non-missing PK assessment.
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms*hours per milliliter
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Micrograms*hours per milliliter
  Trimester 2 (Weeks 18-26 of pregnancy) | 55.045 [37.918 to 79.907]
  Trimester 3 (Weeks 30-36 of pregnancy) | 42.473 [27.613 to 65.330]
  8-12 Weeks postpartum | 78.917 [53.195 to 117.075]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for Dolutegravir
Description: Blood samples were collected at indicated timepoints for PK analysis of dolutegravir at Trimester 2 (Weeks 18-26 of pregnancy), Trimester 3 (Weeks 30-36 of pregnancy) and at 8-12 Weeks postpartum.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms per milliliter
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Micrograms per milliliter
  Trimester 2 (Weeks 18-26 of pregnancy) | 4.420 [2.906 to 6.724]
  Trimester 3 (Weeks 30-36 of pregnancy) | 3.424 [2.038 to 5.753]
  8-12 Weeks Postpartum | 5.578 [3.866 to 8.049]

3. Primary Outcome: Drug Concentration at the End of Dosing Interval (Ctau) for Dolutegravir
Description: as for outcome 2
Time Frame: 24 hours post dose at Trimester 2 (Weeks 18-26 of pregnancy), Trimester 3 (Weeks 30-36 of pregnancy) and at 8-12 Weeks postpartum
Population: Pharmacokinetic Population
Measure: Geometric Mean (95% Confidence Interval); unit: Nanograms per milliliter
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Nanograms per milliliter
  Trimester 2 (Weeks 18-26 of pregnancy) | 930.1 [562.0 to 1539.3]
  Trimester 3 (Weeks 30-36 of pregnancy) | 657.5 [266.1 to 1624.4]
  8-12 Weeks Postpartum | 2154.7 [901.4 to 5150.5]

4. Primary Outcome: Apparent Oral Clearance (CL/F) for Dolutegravir
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (95% Confidence Interval); unit: Liters per hour
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Liters per hour
  Trimester 2 (Weeks 18-26 of pregnancy) | 0.739 [0.484 to 1.130]
  Trimester 3 (Weeks 30-36 of pregnancy) | 0.952 [0.559 to 1.620]
  8-12 Weeks Postpartum | 0.464 [0.062 to 3.476]

5. Primary Outcome: Steady State Volume of Distribution (Vss/F) After Extravascular Administration for Dolutegravir
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (95% Confidence Interval); unit: Liters
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Liters
  Trimester 2 (Weeks 18-26 of pregnancy) | 9.665 [6.651 to 14.044]
  Trimester 3 (Weeks 30-36 of pregnancy) | 12.326 [7.878 to 19.285]
  8-12 Weeks Postpartum | 6.326 [0.048 to 833.336]

6. Primary Outcome: Half-life (T1/2) for Dolutegravir
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Hours
  Trimester 2 (Weeks 18-26 of pregnancy) | 9.215 (1.8968)
  Trimester 3 (Weeks 30-36 of pregnancy) | 9.401 (3.0322)
  8-12 Weeks Postpartum | 9.699 (3.0427)

7. Primary Outcome: Number of Participants (Pregnant Women) With Maximum Severity of Post-Baseline Emergent Hematology Toxicities: Hemoglobin
Description: Blood samples were collected for analysis of hemoglobin. Any abnormality was graded according to Division of Acquired Immunodeficiency Syndrome (DAIDS) toxicity scales from Grade 1 to 4 (1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening). Number of participants (Pregnant Women) with maximum severity of post-Baseline emergent toxicities with respect to hemoglobin has been presented.
Time Frame: Up to Week 32 of study
Population: Safety Population comprised of all participants (Pregnant Women) who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Participants
  Grade 1 | 1
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0

8. Primary Outcome: Absolute Values of the Chemistry Parameters: Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST)
Description: Blood samples were collected for the analysis of chemistry parameters including ALT and AST.
Time Frame: At Baseline (Day 1), Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and Week 32 of study
Population: Safety Population comprised of all participants (Pregnant Women) who received at least one dose of study treatment. Only those participants (pregnant women) with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
International units per Liter
  ALT, Baseline (Day 1), n=4 | 10.8 (5.56)
  ALT, Week 4, n=4 | 15.3 (4.43)
  ALT, Week 8, n=4 | 19.3 (17.21)
  ALT, Week 12, n=4 | 11.0 (3.16)
  ALT, Week 16, n=4 | 10.8 (2.36)
  ALT, Week 20, n=4 | 10.3 (7.27)
  ALT, Week 24, n=1: number analyzed (Participants) | 1
  ALT, Week 24, n=1 | 19.0 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed.
  ALT, Week 32, n=2: number analyzed (Participants) | 2
  ALT, Week 32, n=2 | 28.0 (15.56)
  AST, Baseline (Day 1), n=4 | 14.8 (4.19)
  AST, Week 4, n=4 | 17.3 (2.22)
  AST, Week 8, n=4 | 17.3 (6.18)
  AST, Week 12, n=4 | 15.0 (1.83)
  AST, Week 16, n=4 | 14.8 (2.63)
  AST, Week 20, n=4 | 16.3 (3.30)
  AST, Week 24, n=1: number analyzed (Participants) | 1
  AST, Week 24, n=1 | 20.0 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed.
  AST, Week 32, n=2: number analyzed (Participants) | 2
  AST, Week 32, n=2 | 24.0 (8.49)

9. Primary Outcome: Change From Baseline in Chemistry Parameters: ALT and AST
Description: Blood samples were collected for the analysis of chemistry parameters including ALT and AST. Baseline value (Day 1) is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and Week 32 of study
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
International units per Liter
  ALT, Week 4, n=4 | 4.5 (6.03)
  ALT, Week 8, n=4 | 8.5 (11.79)
  ALT, Week 12, n=4 | 0.3 (3.30)
  ALT, Week 16, n=4 | 0.0 (3.56)
  ALT, Week 20, n=4 | -0.5 (1.73)
  ALT, Week 24, n=1: number analyzed (Participants) | 1
  ALT, Week 24, n=1 | 0.0 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed.
  ALT, Week 32, n=2: number analyzed (Participants) | 2
  ALT, Week 32, n=2 | 19.5 (14.85)
  AST, Week 4, n=4 | 2.5 (4.43)
  AST, Week 8, n=4 | 2.5 (2.38)
  AST, Week 12, n=4 | 0.3 (3.10)
  AST, Week 16, n=4 | 0.0 (3.37)
  AST, Week 20, n=4 | 1.5 (1.29)
  AST, Week 24, n=1: number analyzed (Participants) | 1
  AST, Week 24, n=1 | -1.0 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed.
  AST, Week 32, n=2: number analyzed (Participants) | 2
  AST, Week 32, n=2 | 11.0 (8.49)

10. Primary Outcome: Absolute Values of the Chemistry Parameters: Bilirubin and Creatinine
Description: Blood samples were collected for the analysis of chemistry parameters including Bilirubin and Creatinine.
Time Frame: At Baseline (Day 1), Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and Week 32 of study
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Micromoles per Liter
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Micromoles per Liter
  Bilirubin, Baseline (Day 1), n=4 | 7.3 (3.77)
  Bilirubin, Week 4, n=4 | 5.0 (1.83)
  Bilirubin, Week 8, n=4 | 5.5 (2.65)
  Bilirubin, Week 12, n=4 | 4.5 (1.29)
  Bilirubin, Week 16, n=4 | 4.5 (1.29)
  Bilirubin, Week 20, n=4 | 4.5 (1.29)
  Bilirubin, Week 24, n=1: number analyzed (Participants) | 1
  Bilirubin, Week 24, n=1 | 7.0 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed.
  Bilirubin, Week 32, n=2: number analyzed (Participants) | 2
  Bilirubin, Week 32, n=2 | 6.5 (0.71)
  Creatinine, Baseline (Day 1), n=4 | 57.73 (16.661)
  Creatinine, Week 4, n=4 | 50.50 (2.990)
  Creatinine, Week 8, n=4 | 51.58 (3.067)
  Creatinine, Week 12, n=4 | 50.68 (3.293)
  Creatinine, Week 16, n=4 | 47.45 (2.001)
  Creatinine, Week 20, n=4 | 50.60 (6.424)
  Creatinine, Week 24, n=1: number analyzed (Participants) | 1
  Creatinine, Week 24, n=1 | 63.60 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed.
  Creatinine, Week 32, n=2: number analyzed (Participants) | 2
  Creatinine, Week 32, n=2 | 68.90 (3.677)

11. Primary Outcome: Change From Baseline in Chemistry Parameters: Bilirubin and Creatinine
Description: Blood samples were collected for the analysis of chemistry parameters including Bilirubin and Creatinine. Baseline value (Day 1) is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and Week 32 of study
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Micromoles per Liter
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Micromoles per Liter
  Bilirubin, Week 4, n=4 | -2.3 (2.06)
  Bilirubin, Week 8, n=4 | -1.8 (1.26)
  Bilirubin, Week 12, n=4 | -2.8 (2.99)
  Bilirubin, Week 16, n=4 | -2.8 (2.99)
  Bilirubin, Week 20, n=4 | -2.8 (2.99)
  Bilirubin, Week 24, n=1: number analyzed (Participants) | 1
  Bilirubin, Week 24, n=1 | -5.0 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed.
  Bilirubin, Week 32, n=2: number analyzed (Participants) | 2
  Bilirubin, Week 32, n=2 | 2.0 (2.83)
  Creatinine, Week 4, n=4 | -7.23 (14.014)
  Creatinine, Week 8, n=4 | -6.15 (16.700)
  Creatinine, Week 12, n=4 | -7.05 (14.328)
  Creatinine, Week 16, n=4 | -10.28 (17.453)
  Creatinine, Week 20, n=4 | -7.13 (11.154)
  Creatinine, Week 24, n=1: number analyzed (Participants) | 1
  Creatinine, Week 24, n=1 | -19.10 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed.
  Creatinine, Week 32, n=2: number analyzed (Participants) | 2
  Creatinine, Week 32, n=2 | 19.10 (3.253)

12. Primary Outcome: Absolute Values of the Hematology Parameters: Hemoglobin
Description: Blood samples were collected for the analysis of hematology parameters including hemoglobin.
Time Frame: At Baseline (Day 1), Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and Week 32 of study
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Grams per Liter
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Grams per Liter
  Baseline (Day 1), n=4 | 127.8 (11.24)
  Week 4, n=4 | 120.8 (7.23)
  Week 8, n=4 | 113.5 (7.05)
  Week 12, n=4 | 116.5 (7.14)
  Week 16, n=4 | 115.0 (4.69)
  Week 20, n=4 | 115.8 (8.30)
  Week 24, n=1: number analyzed (Participants) | 1
  Week 24, n=1 | 127.0 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed.
  Week 32, n=2: number analyzed (Participants) | 2
  Week 32, n=2 | 140.5 (0.71)

13. Primary Outcome: Change From Baseline in Hematology Parameters: Hemoglobin
Description: Blood samples were collected for the analysis of hematology parameters including hemoglobin. Baseline value (Day 1) is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and Week 32 of study
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Grams per Liter
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Grams per Liter
  Week 4, n=4 | -7.0 (10.17)
  Week 8, n=4 | -14.3 (7.37)
  Week 12, n=4 | -11.3 (4.92)
  Week 16, n=4 | -12.8 (6.65)
  Week 20, n=4 | -12.0 (4.97)
  Week 24, n=1: number analyzed (Participants) | 1
  Week 24, n=1 | -14.0 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed.
  Week 32, n=2: number analyzed (Participants) | 2
  Week 32, n=2 | 14.0 (8.49)

14. Primary Outcome: Absolute Values of the Hematology Parameters: Leukocytes and Platelets
Description: Blood samples were collected for the analysis of hematology parameters including leukocytes and platelets.
Time Frame: At Baseline (Day 1), Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and Week 32 of study
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Giga cells per Liter
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Giga cells per Liter
  Leukocytes, Baseline (Day 1), n=4 | 6.48 (1.415)
  Leukocytes, Week 4, n=4 | 7.88 (2.095)
  Leukocytes, Week 8, n=4 | 8.43 (1.959)
  Leukocytes, Week 12, n=4 | 9.15 (2.053)
  Leukocytes, Week 16, n=4 | 9.23 (1.821)
  Leukocytes, Week 20, n=4 | 10.03 (2.848)
  Leukocytes, Week 24, n=1: number analyzed (Participants) | 1
  Leukocytes, Week 24, n=1 | 12.60 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed.
  Leukocytes, Week 32, n=2: number analyzed (Participants) | 2
  Leukocytes, Week 32, n=2 | 5.85 (0.636)
  Platelets, Baseline (Day 1), n=4 | 204.8 (37.03)
  Platelets, Week 4, n=4 | 200.5 (2.38)
  Platelets, Week 8, n=4 | 220.8 (16.07)
  Platelets, Week 12, n=4 | 195.5 (25.38)
  Platelets, Week 16, n=4 | 198.0 (10.80)
  Platelets, Week 20, n=4 | 216.5 (10.91)
  Platelets, Week 24, n=1: number analyzed (Participants) | 1
  Platelets, Week 24, n=1 | 250.0 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed.
  Platelets, Week 32, n=2: number analyzed (Participants) | 2
  Platelets, Week 32, n=2 | 206.0 (24.04)

15. Primary Outcome: Change From Baseline in Hematology Parameters: Leukocytes and Platelets
Description: Blood samples were collected for the analysis of hematology parameters including leukocytes and platelets. Baseline value (Day 1) is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and Week 32 of study
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Giga cells per Liter
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Giga cells per Liter
  Leukocytes, Week 4, n=4 | 1.40 (1.817)
  Leukocytes, Week 8, n=4 | 1.95 (2.047)
  Leukocytes, Week 12, n=4 | 2.68 (1.173)
  Leukocytes, Week 16, n=4 | 2.75 (1.654)
  Leukocytes, Week 20, n=4 | 3.55 (2.340)
  Leukocytes, Week 24, n=1: number analyzed (Participants) | 1
  Leukocytes, Week 24, n=1 | 4.90 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed.
  Leukocytes, Week 32, n=2: number analyzed (Participants) | 2
  Leukocytes, Week 32, n=2 | -0.65 (1.061)
  Platelets, Week 4, n=4 | -4.3 (39.09)
  Platelets, Week 8, n=4 | 16.0 (33.44)
  Platelets, Week 12, n=4 | -9.3 (39.08)
  Platelets, Week 16, n=4 | -6.8 (47.16)
  Platelets, Week 20, n=4 | 11.8 (45.49)
  Platelets, Week 24, n=1: number analyzed (Participants) | 1
  Platelets, Week 24, n=1 | 10.0 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed.
  Platelets, Week 32, n=2: number analyzed (Participants) | 2
  Platelets, Week 32, n=2 | -4.0 (50.91)

16. Primary Outcome: Number of Participants (Pregnant Women) Who Discontinued the Treatment Due to Adverse Events (AE)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a study treatment. Number of participants (pregnant women) who discontinued the treatment due to adverse events have been presented.
Time Frame: Up to Week 292
Population: Safety Population comprised of all participants (Pregnant Women) who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Participants | 0

17. Primary Outcome: Number of Participants (Pregnant Women) Demonstrated Congenital Malformations
Description: Data for participants (pregnant women) demonstrated congenital malformations was reported.
Time Frame: At delivery (up to Week 40 of pregnancy)
Population: Safety Population comprised of all participants (Pregnant Women) who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Participants | 0

18. Secondary Outcome: Time to Cmax (Tmax) for Dolutegravir
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Hours
  Trimester 2 (Weeks 18-26 of pregnancy) | 3.508 (1.7082)
  Trimester 3 (Weeks 30-36 of pregnancy) | 2.729 (0.4877)
  8-12 Weeks Postpartum | 4.242 (2.0522)

19. Secondary Outcome: Pre-dose Plasma Concentration (C0) for Dolutegravir
Description: as for outcome 2
Time Frame: Pre-dose at Trimester 2 (Weeks 18-26 of pregnancy), Trimester 3 (Weeks 30-36 of pregnancy) and at 8-12 Weeks postpartum
Population: Pharmacokinetic Population
Measure: Geometric Mean (95% Confidence Interval); unit: Nanograms per milliliter
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Nanograms per milliliter
  Trimester 2 (Weeks 18-26 of pregnancy) | 666.9 [149.5 to 2974.6]
  Trimester 3 (Weeks 30-36 of pregnancy) | 1084.6 [676.7 to 1738.3]
  8-12 Weeks Postpartum | 1225.0 [522.8 to 2870.1]

20. Secondary Outcome: Unbound DTG Concentrations in Plasma at 3 and 24 Hours Post Dose of Dolutegravir
Description: as for outcome 2
Time Frame: At 3 hours and 24 hours post dose in Trimester 2 (Weeks 18-26 of pregnancy), Trimester 3 (Weeks 30-36 of pregnancy) and at 8-12 Weeks postpartum
Population: Pharmacokinetic Population
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms per milliliter
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Micrograms per milliliter
  At 3 hours post dose in Trimester 2 | 7.856 [4.370 to 14.122]
  At 3 hours post dose in Trimester 3 | 7.371 [4.594 to 11.827]
  At 3 hours post dose 8-12 Weeks postpartum | 6.898 [4.360 to 10.914]
  At 24 hours post dose in Trimester 2 | 1.798 [0.887 to 3.644]
  At 24 hours post dose in Trimester 3 | 2.065 [1.229 to 3.471]
  At 24 hours post dose 8-12 Weeks postpartum | 2.881 [1.503 to 5.520]

21. Secondary Outcome: Total DTG Concentrations in Plasma From Cord Blood and Maternal Blood at the Time of Delivery
Description: Blood samples were collected at the time of delivery for PK analysis of dolutegravir.
Time Frame: At delivery (up to Week 40 of pregnancy)
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Nanograms per milliliter
  Cord plasma concentration | 1436.0 (1287.43)
  Maternal plasma concentration | 1806.3 (1125.04)

22. Secondary Outcome: Number of Participants (Pregnant Women) With Treatment-emergent Genotypic and/or Phenotypic Resistance Who Met Confirmed Virologic Withdrawal Criteria
Description: Number of participants (pregnant women) with treatment-emergent genotypic and/or phenotypic resistance who met confirmed virologic withdrawal criteria are presented. Genotypic and phenotypic analyses were carried out by Monogram Biosciences using, but not limited to, their Standard Phenosense and GenoSure testing methods for protease (PRO) and reverse transcriptase (RT), or with their GeneSeq Integrase and PhenoSense Integrase assays.
Time Frame: Up to Week 32 of study
Population: Intent-to-Treat Exposed (ITT-E) Population includes all participants (pregnant women) who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Participants
  Participants with genotypic resistance | 0
  Participants with phenotypic resistance | 0

23. Secondary Outcome: Number of Participants (Pregnant Women) With Live Birth Outcome Categories
Description: Participants (pregnant women) with following live birth outcome categories are reported- Vaginal Birth, Planned Caesarean Section, Unscheduled Caesarean Section and Preterm Delivery.
Time Frame: At delivery (up to Week 40 of pregnancy)
Population: Safety Population comprised of all participants (Pregnant Women) who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Participants
  Vaginal Birth | 1
  Planned Caesarean Section | 2
  Unscheduled Caesarean Section | 1
  Preterm Delivery | 1

24. Secondary Outcome: Gestational Age of Infants
Description: Gestational age is defined as the number of weeks between the first day of the mother's last normal menstrual period and the day of birth. Data for gestational age of infants has been presented.
Time Frame: At birth
Population: Analysis was performed on Infant Population which consisted of infants born to pregnant women who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: Weeks
Groups:
- DTG/ABC/3TC - Infant: This group consisted of Infants born to pregnant women who received a fixed dose combination tablet of dolutegravir, abacavir and lamivudine during pregnancy.
Arm/Group | DTG/ABC/3TC - Infant
Number analyzed (Participants) | 4
Weeks | 38.3 (1.71)

25. Secondary Outcome: Neonatal Length and Head Circumference at Birth
Description: Data for neonatal length and head circumference at birth are reported.
Time Frame: At birth
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | DTG/ABC/3TC - Infant
Number analyzed (Participants) | 4
Centimeter
  Neonatal Length | 51.5 (3.11)
  Neonatal Head Circumference | 34.9 (1.65)

26. Secondary Outcome: Neonatal Weight at Birth
Description: Data for neonatal weight at birth has been reported.
Time Frame: At birth
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | DTG/ABC/3TC - Infant
Number analyzed (Participants) | 4
Grams | 3262.5 (731.36)

27. Secondary Outcome: Number of Infants by Their Weight Categories at Birth
Description: Weight of infants at birth were categorized as: Small for Gestational Age (SGA) defined neonates under the 10th percentile in weight, Appropriate for Gestational Age (AGA) characterized neonates between the 10th and 90th percentiles in weight and Large for Gestational Age (LGA) referred to neonates over the 90th percentile in weight.
Time Frame: At birth
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/ABC/3TC - Infant
Number analyzed (Participants) | 4
Participants
  LGA | 0
  AGA | 4
  SGA | 0

28. Secondary Outcome: Number of Infants by Appearance, Pulse, Grimace, Activity, and Respiration (APGAR) Score at 1 and 5 Minutes After Birth
Description: APGAR is a quick test to assess the health of new born. The test is performed at 1 and 5 minutes after birth. APGAR scale is determined by evaluating the new born on five categories (appearance, pulse, grimace, activity and respiration) on a scale from zero to two with 2 being the best score, then summing up the values obtained from all five categories. APGAR score ranges from 0 to 10 (Higher score indicates better health) where a score of 7 and above is normal. Number of infants by APGAR score at 1 and 5 minutes after birth are presented.
Time Frame: 1 and 5 minutes after birth
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/ABC/3TC - Infant
Number analyzed (Participants) | 4
Participants
  1 Minute, Score 0 to 6 | 0
  1 Minute, Score 7 to 10 | 4
  5 Minute, Score 0 to 6 | 0
  5 Minute, Score 7 to 10 | 4

29. Secondary Outcome: Percentage of Participants (Pregnant Women) With Plasma Human Immunodeficiency Virus Type 1 (HIV-1) Ribonucleic Acid (RNA) <50 Copies/Milliliter (c/mL) by Visit
Description: Percentage of participants (pregnant women) with plasma HIV-1 RNA <50 c/mL are presented. Plasma samples were collected for quantitative analysis of HIV-1 RNA.
Time Frame: At Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28 and Week 32 of study
Population: Intent-to-Treat Exposed Population. Only those participants (pregnant women) with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Number; unit: Percentage of participants
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Percentage of participants
  Week 4, n=4 | 100
  Week 8, n=4 | 100
  Week 12, n=4 | 100
  Week 16, n=4 | 100
  Week 20, n=4 | 100
  Week 24, n=2: number analyzed (Participants) | 2
  Week 24, n=2 | 100
  Week 28, n=1: number analyzed (Participants) | 1
  Week 28, n=1 | 100
  Week 32, n=2: number analyzed (Participants) | 2
  Week 32, n=2 | 100

30. Secondary Outcome: Percentage of Participants (Pregnant Women) With Plasma HIV-1 RNA <400 c/mL by Visit
Description: Percentage of participants (pregnant women) with plasma HIV-1 RNA <400 c/mL are presented. Plasma samples were collected for quantitative analysis of HIV-1 RNA.
Time Frame: At Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28 and Week 32 of study
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Percentage of participants
  Week 4, n=4 | 100
  Week 8, n=4 | 100
  Week 12, n=4 | 100
  Week 16, n=4 | 100
  Week 20, n=4 | 100
  Week 24, n=2: number analyzed (Participants) | 2
  Week 24, n=2 | 100
  Week 28, n=1: number analyzed (Participants) | 1
  Week 28, n=1 | 100
  Week 32, n=2: number analyzed (Participants) | 2
  Week 32, n=2 | 100

31. Secondary Outcome: Absolute Values of Cluster of Differentiation 4 (CD4+) T Cell Counts by Visit
Description: Blood samples were collected for the analysis of CD4+ T cell counts using cytometry.
Time Frame: At Baseline (Day 1), Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28 and Week 32 of study
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Cells per cubic millimeter
  Baseline (Day 1), n=4 | 476.3 (123.31)
  Week 4, n=4 | 569.5 (238.51)
  Week 8, n=4 | 569.8 (296.43)
  Week 12, n=4 | 575.0 (331.22)
  Week 16, n=4 | 626.8 (270.63)
  Week 20, n=4 | 791.5 (524.96)
  Week 24, n=2: number analyzed (Participants) | 2
  Week 24, n=2 | 874.5 (516.90)
  Week 28, n=1: number analyzed (Participants) | 1
  Week 28, n=1 | 488.0 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed.
  Week 32, n=2: number analyzed (Participants) | 2
  Week 32, n=2 | 677.5 (40.31)

32. Secondary Outcome: Change From Baseline in CD4+ T Cell Counts by Visit
Description: Blood samples were collected for the analysis of CD4+ T cell counts using cytometry. Baseline value (Day 1) is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28 and Week 32 of study
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Cells per cubic millimeter
  Week 4, n=4 | 93.3 (124.64)
  Week 8, n=4 | 93.5 (174.54)
  Week 12, n=4 | 98.8 (208.50)
  Week 16, n=4 | 150.5 (148.73)
  Week 20, n=4 | 315.3 (402.00)
  Week 24, n=2: number analyzed (Participants) | 2
  Week 24, n=2 | 353.0 (332.34)
  Week 28, n=1: number analyzed (Participants) | 1
  Week 28, n=1 | 98.0 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed.
  Week 32, n=2: number analyzed (Participants) | 2
  Week 32, n=2 | 246.0 (97.58)

33. Secondary Outcome: Number of Participants (Pregnant Women) With Disease Progression
Description: Disease progression included HIV-associated conditions, acquired immunodeficiency syndrome (AIDS) and death. Number of participants (pregnant women) with disease progression to Centers for Disease Control and Prevention (CDC) class C or death have been presented.
Time Frame: Up to Week 32 of study
Population: Intent-to-Treat Exposed Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Participants | 0

34. Primary Outcome: Number of Participants (Pregnant Women) With Adverse Events (AE) as Per Severity Grades
Description: Number of participants (pregnant women) with adverse events (AE) as per severity grades were presented. Grade 1 is mild, grade 2 is moderate, grade 3 is severe or medically significant but not immediately life-threatening and grade 4 is life-threatening consequences; urgent intervention required.
Time Frame: Up to 292 Weeks
Population: Safety Population comprised of all participants (Pregnant Women) who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/ABC/3TC - Mother
Number analyzed (Participants) | 4
Participants
  Grade 1 | 2
  Grade 2 | 2
  Grade 3 | 0
  Grade 4 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events (SAEs) and non-serious adverse events (non-SAEs) were collected up to Week 328
Description: Safety population comprised of all pregnant women who received at least one dose of study treatment. All-Cause Mortality, SAEs and non-SAEs were collected only in pregnant women (enrolled population/study participants) and not in infants, as infants were not considered as enrolled per study design.
Arm/Group | DTG/ABC/3TC - Mother | DTG/ABC/3TC - Infant
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/0
Other Adverse Events (participants affected / at risk) | 4/4 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG/ABC/3TC - Mother (N=4) | DTG/ABC/3TC - Infant (N=0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG/ABC/3TC - Mother (N=4) | DTG/ABC/3TC - Infant (N=0)
Respiratory tract infection (Infections and infestations) | 2 (5) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 1 (2) | 0 (0)
Nephropathy (Renal and urinary disorders) | 2 (4) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT02075593/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT02075593/SAP_002.pdf